CLINICAL TRIAL: NCT06473246
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Study to Determine Safety, Pharmakokinetics and Efficacy of the Different Doses of VL-SE-01 in Healthy Participants.
Brief Title: A Study to Determine Safety, Pharmakokinetics and Efficacy of the Different Doses of VL-SE-01 in Healthy Participants.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SE/230302/CBD/SS
Record Dates: First submitted 2024-06-03; First posted 2024-06-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy Population

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind and Placebo controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CBD Isolate (25 mg/0.5 ml) (Active Comparator): 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Interventions: Dietary Supplement: CBD Isolate (25 mg/0.5 ml)
- CBD Isolate (40 mg/0.5 ml) (Active Comparator): 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Interventions: Dietary Supplement: CBD Isolate (40 mg/0.5 ml)
- CBD Isolate (50 mg/0.5 ml) (Active Comparator): 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Interventions: Dietary Supplement: CBD Isolate (50 mg/0.5 ml)
- CBD Broad Extract (50 mg/0.5 ml) (Active Comparator): 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Interventions: Dietary Supplement: CBD Broad Extract (50 mg/0.5 ml)
- Placebo (Placebo Comparator): 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CBD Isolate (25 mg/0.5 ml) — 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Arms: CBD Isolate (25 mg/0.5 ml)
Dietary Supplement: CBD Isolate (40 mg/0.5 ml) — 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Arms: CBD Isolate (40 mg/0.5 ml)
Dietary Supplement: CBD Isolate (50 mg/0.5 ml) — 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Arms: CBD Isolate (50 mg/0.5 ml)
Dietary Supplement: CBD Broad Extract (50 mg/0.5 ml) — 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Arms: CBD Broad Extract (50 mg/0.5 ml)
Dietary Supplement: Placebo — 0.5 ml sublingually to be consumed after dinner, 30 min ± 5 mins before going to bed.
  Arms: Placebo

SUMMARY:
The present study is a randomized, placebo-controlled, parallel study. 250 participants will be screened, and considering a screening failure rate of 20%, approximately 200 participants will be randomized in a ratio of 1:1:1:1:1 to receive either different doses of VL-SE-01 or placebo and will be assigned a unique randomization code. Each group will have at least 30 participants (total 150 completers) after accounting for a dropout/withdrawal rate of 25%. The intervention duration for all the study participants is 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Male & female individuals must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Individuals who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Individual has a body weight of at least 50 kg (males) or 45 kg (females) and body mass index (BMI) within the range 18.5 to 29.9 kg/m2 (inclusive)
* Individuals with a stressed lifestyle as assessed by PSS scores within 27- 40.
* A male must agree to use contraception during the intervention period and for at least 7 days after the last dose of study intervention and refrain from donating sperm during this period.
* A female is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP)
  2. OR agrees to use the contraceptive during the intervention period and for at least 90 days after the last dose of study intervention

Exclusion Criteria:

* Individual has a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinology related, haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention, or interfering with the interpretation of data.
* Males who has a history of oligospermia, vasectomy and other sperm abnormalities.
* Females who have irregularity or problems in menstrual cycles or diagnosed with polycystic ovarian syndrome.
* Individuals with Type 1 and Type 2 Diabetes mellitus and on medication.
* Individuals with SBP ≥ 160 mmHg and DBP ≥ 100 mmHg.
* Individuals on anti-hypertensives.
* History and/or current cases of chronic alcohol consumption or heavy drinkers as defined by:

  1. For men, consuming more than 4 drinks on any day or more than 14 drinks/week
  2. For women, consuming more than 3 drinks on any day or more than 7 drinks/week
* Peri and post-menopausal women with no menstrual cycle in the last 6 months
* Individuals with a history or actively under the influence of Hemp or CBD products by any means of administration
* Individual has a known hypersensitivity to any components of the study medication or comparative drugs (and/or an investigational device) as stated in this protocol
* Individual has a history of unexplained syncope or a family history of sudden death due to long QT syndrome
* Individual with a history and/or currently diagnosed of cancer like lymphoma, leukaemia, or any malignancy.
* Individual has past or intended use of prohibited medication or prescription medication including herbal medications within 2 weeks or 5 half-lives prior to dosing
* Individuals have taken sleep medication within 2 weeks prior to screening
* Individual has used hepatic enzyme-inducing drugs within 2 months prior to dosing
* Individuals has alanine transaminase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.5 times upper limit of normal (ULN)
* Individual has current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Individual has any clinically relevant electrocardiogram (ECG) finding at the Screening Visit or at Baseline
* Individual has a history of human immunodeficiency virus (HIV), hepatitis B, and hepatitis C.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of VL-SE-01 by assessing Fasting Blood Glucose as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day -5 to Day -1
  Fasting Glucose normal range is 74 - 106 mg/dL
To evaluate the safety of VL-SE-01 by assessing Fasting Blood Glucose as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day 90
  Fasting Glucose normal range is 74 - 106 mg/dL
To evaluate the safety of VL-SE-01 by assessing Fasting Blood Glucose as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day 180
  Fasting Glucose normal range is 74 - 106 mg/dL
To evaluate the safety of VL-SE-01 by assessing Renal function as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day -5 to Day -1
  Renal function tests measure the efficiency of kidneys and include Electrolytes (Sodium, Potassium, and Chloride), Creatinine, Glomerular Filtration Rate (GFR), Blood Urea Nitrogen, Blood Urea and Calcium tests.
  Normal range for these tests are mentioned below:
  Sodium:136 - 145 mmol/L Potassium: 3.5 - 5.1 mmol/L Chloride: 98 - 107 mmol/L Creatinine: Males - 0.7 - 1.2 mg/dL; Females - 0.5 - 0.9 mg/dL
  GFR:
  Blood Urea Nitrogen: Males - 18 yrs - 49 yrs : 8.87-22.88 mg/dL, > 50 yrs : 9.80-22.88 mg/dL; Females - 18 yrs - 49 yrs : 7.47-17.74 mg/dL, > 50 yrs : 8.87-21.94 mg/dL Blood Urea: Males - 18 yrs - 49 yrs : 19 - 49 mg/dL, > 50 yrs : 21 - 49 mg/dL; Females - 18 yrs - 49 yrs : 16 - 38 mg/dL, > 50 yrs : 19 - 47 mg/dL Calcium: 8.6 - 10.0 mg/dL
To evaluate the safety of VL-SE-01 by assessing Renal function as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day 90
  Renal function tests measure the efficiency of kidneys and include Electrolytes (Sodium, Potassium, and Chloride), Creatinine, Glomerular Filtration Rate (GFR), Blood Urea Nitrogen, Blood Urea and Calcium tests.
  Normal range for these tests are mentioned below:
  Sodium:136 - 145 mmol/L Potassium: 3.5 - 5.1 mmol/L Chloride: 98 - 107 mmol/L Creatinine: Males - 0.7 - 1.2 mg/dL; Females - 0.5 - 0.9 mg/dL
  GFR:
  Blood Urea Nitrogen: Males - 18 yrs - 49 yrs : 8.87-22.88 mg/dL, > 50 yrs : 9.80-22.88 mg/dL; Females - 18 yrs - 49 yrs : 7.47-17.74 mg/dL, > 50 yrs : 8.87-21.94 mg/dL Blood Urea: Males - 18 yrs - 49 yrs : 19 - 49 mg/dL, > 50 yrs : 21 - 49 mg/dL; Females - 18 yrs - 49 yrs : 16 - 38 mg/dL, > 50 yrs : 19 - 47 mg/dL Calcium: 8.6 - 10.0 mg/dL
To evaluate the safety of VL-SE-01 by assessing Renal function as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day 180
  Renal function tests measure the efficiency of kidneys and include Electrolytes (Sodium, Potassium, and Chloride), Creatinine, Estimated Glomerular Filtration Rate (eGFR), Blood Urea Nitrogen, Blood Urea and Calcium tests.
  Normal range for these tests are mentioned below:
  Sodium:136 - 145 mmol/L Potassium: 3.5 - 5.1 mmol/L Chloride: 98 - 107 mmol/L Creatinine: Males - 0.7 - 1.2 mg/dL; Females - 0.5 - 0.9 mg/dL eGFR: 60 - 200 mL/min/1.73 m² Blood Urea Nitrogen: Males - 18 yrs - 49 yrs : 8.87-22.88 mg/dL, > 50 yrs : 9.80-22.88 mg/dL; Females - 18 yrs - 49 yrs : 7.47-17.74 mg/dL, > 50 yrs : 8.87-21.94 mg/dL Blood Urea: Males - 18 yrs - 49 yrs : 19 - 49 mg/dL, > 50 yrs : 21 - 49 mg/dL; Females - 18 yrs - 49 yrs : 16 - 38 mg/dL, > 50 yrs : 19 - 47 mg/dL Calcium: 8.6 - 10.0 mg/dL
To evaluate the safety of VL-SE-01 by assessing Liver function as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day -5 to -1
  Liver Function tests help determine the health of liver by measuring the levels of Albumin, Total Proteins, Alkaline Phosphatase (ALP), Alanine transaminase (ALT), Aspartate aminotransferase (AST), Bilirubin, and gamma-glutamyl transferase (GGT) levels in blood.
  Albumin: 3.5 - 5.2 g/dL Total Proteins: 6.6 - 8.9 g/dL Alkaline Phosphatase: Males - 40 - 129 U/L; Females - 35 - 104 U/L ALT: Males - Up to 41 U/L; Females - Up to 33 U/L AST: Males - Up to 40 U/L; Females - Up to 32 U/L Bilirubin: Total Bilirubin - Up to 1.2 mg/dL; Direct Bilirubin - Up to 0.3 mg/dL; Indirect Bilirubin - Up to 0.9 mg/dL GGT: Males - 10 - 71 U/L; Females - 6 - 42 U/L
To evaluate the safety of VL-SE-01 by assessing Liver function as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day 90
  Liver Function tests help determine the health of liver by measuring the levels of Albumin, Total Proteins, Alkaline Phosphatase (ALP), Alanine transaminase (ALT), Aspartate aminotransferase (AST), Bilirubin, and gamma-glutamyl transferase (GGT) levels in blood.
  Albumin: 3.5 - 5.2 g/dL Total Proteins: 6.6 - 8.9 g/dL Alkaline Phosphatase: Males - 40 - 129 U/L; Females - 35 - 104 U/L ALT: Males - Up to 41 U/L; Females - Up to 33 U/L AST: Males - Up to 40 U/L; Females - Up to 32 U/L Bilirubin: Total Bilirubin - Up to 1.2 mg/dL; Direct Bilirubin - Up to 0.3 mg/dL; Indirect Bilirubin - Up to 0.9 mg/dL GGT: Males - 10 - 71 U/L; Females - 6 - 42 U/L
To evaluate the safety of VL-SE-01 by assessing Liver function as part of the Complete Metabolic Panel (CMP) before and after IP consumption. | Day 180
  Liver Function tests help determine the health of liver by measuring the levels of Albumin, Total Proteins, Alkaline Phosphatase (ALP), Alanine transaminase (ALT), Aspartate aminotransferase (AST), Bilirubin, and gamma-glutamyl transferase (GGT) levels in blood.
  Albumin: 3.5 - 5.2 g/dL Total Proteins: 6.6 - 8.9 g/dL Alkaline Phosphatase: Males - 40 - 129 U/L; Females - 35 - 104 U/L ALT: Males - Up to 41 U/L; Females - Up to 33 U/L AST: Males - Up to 40 U/L; Females - Up to 32 U/L Bilirubin: Total Bilirubin - Up to 1.2 mg/dL; Direct Bilirubin - Up to 0.3 mg/dL; Indirect Bilirubin - Up to 0.9 mg/dL GGT: Males - 10 - 71 U/L; Females - 6 - 42 U/L

SECONDARY OUTCOMES:
To assess the safety and tolerability of VL-SE-01 using blood, which includes Complete Blood Count (CBC). | Day -5 to Day -1, Day 90, Day 180 and Day 195
  CBC measures red blood cells (RBC) which basically carries oxygen, white blood cells (WBC)(Leukocytes), which fights with infection, hemoglobin (Hb), which carries oxygen protein in blood cells, and platelets, which help blood to clot. A complete blood count can show unusual increases or decreases in cell counts.
  Normal ranges for the parameters are as follows:
  Hb: Males: 13 - 17 g/dL; Females - 11.5 - 15.2 g/dL Total RBC: Males - 4.2 - 6.0 million cells/cumm; Females - 3.8 - 5.2 million cells/cumm Total WBC: 3500 - 10000 / cumm Platelet Count: 150000 - 400000 / cumm
To assess the safety and tolerability of VL-SE-01 using blood, which includes Inflammation by analyzing CRP levels. | Day 0, Day 90, Day 180 and Day 195
  Normal reference range: 0 -5.0 mg/L
To assess the safety and tolerability of VL-SE-01 using blood, which includes Hormonal profile (Luteinizing hormone (LH), follicle-stimulating hormone (FSH), testosterone, estradiol and progesterone) | Day 0, Day 90, Day 180 and Day 195
  Leutinizing Hormone in Females reference range:
  Follicular Phase : 2.4 - 12.6 mIU/mL Ovulating Phase : 14.0 - 95.6 mIU/mL Luteal Phase : 1.0 - 11.4 mIU/mL Post menopausal : 7.7 - 58.5 mIU/mL
  Follicular Stimulating Hormones in Females reference range:
  Follicular Phase : 3.5 - 12.5 mIU/mL Ovulating Phase : 4.7 - 21.5 mIU/mL Luteal Phase : 1.7 - 7.7 mIU/mL Post menopausal : 25.8 - 134.8 mIU/mL
  Progesterone in Females reference ranges:
  Follicular phase: 0.2 - 1.5 ng/ml Ovulatory phase: 0.8 - 3.0 ng/ml Luteal phase: 1.7 - 27.0 ng/ml Post menopause: 0.1 - 0.8 ng/ml
  Estradiol in females reference range:
  Follicular phase :12.5-166 pg/ml Ovulatory phase :85.5-498 pg/ml Luteal phase : 43.8-211 pg/ml Post menopause : 5.0-54.7 pg/ml Pregnancy,1st trimester: 215-4300 pg/ml
  Testosterone in Males reference range: 2.8 - 8.0 ng/mL
To assess the safety and tolerability of VL-SE-01 using blood, which includes Thyroid profile (T3, T4, TSH) | Day 0, Day 90, Day 180 and Day 195
  Total Triiodothyronine (T3) reference range: 1.3 - 3.1 nmol/L Total Thyroxine (T4) reference range: 5.1 - 14.1 μg/dL Thyroid Stimulating Hormone (TSH) reference range: 0.27 - 4.2 μIU/mL
To assess the safety and tolerability of VL-SE-01 using blood, which includes Lipid Profile as assessed by levels of total cholesterol, LDL, HDL and triglycerides | Day 0, Day 90, Day 180 and Day 195
  Total Cholesterol: Desirable: < 200 mg/dL, Borderline High : 200 - 239 mg/dL, High : ≥ 240 mg/dL Triglyceride: Normal : < 150 mg/dL, Borderline : 151 - 199 mg/dL, High : 200 - 499 mg/dL, Very High : > 500 mg/dL HDL Cholesterol: 40 - 60 mg/dL LDL Cholesterol: Optimal : < 100 mg/dL, Near / Above Optimal : 101-129 mg/dL, Borderline High : 130 - 159 mg/dL, High : 160 -189 mg/dL, Very High : > 190 mg/dL
To assess the safety and tolerability of VL-SE-01 on Semen. | Day -5 to Day -1 and Day 180
  Assessment of semen will be done using the following parameters:
  Physical examination which includes factors like Volume (>1.5 ml), appearance, Colour, Viscosity (<2 cm thread after liquefaction) and pH (>= 7.2) of the sample.
  Microscopic Examination which includes Sperm count [Sperm concentration is the number of sperm per milliliter of semen (Reference Range: >=16 Million/ml)] and Motility [Sperm motility is the ability of your sperm to swim (>=42 %)]
To assess the safety and tolerability of VL-SE-01 using blood Plasma levels of CBD and its metabolites [7-Carboxy-cannabidiol (7-COOH-CBD) and 7-Hydroxy-cannabidiol (7-OH-CBD)] | Day 195 (single timepoint)
  (will be conducted in 15 participants only in each group except placebo)
To assess the safety and tolerability of VL-SE-01 on Blood Pressure. | Day 0, Day 90, Day 180 and Day 195
  Vitals signs measures basic functions of the body. In this case, Blood pressure (BP) will be measured.
  Blood pressure will be measured using a calibrated digital monitor.
  Systolic BP (measured in mmHg): Optimal - <120, Normal - 120 - 129, High normal - 130 - 139, Grade 1 hypertension - 140 - 159, Grade 2 hypertension - 160 - 179, Grade 3 hypertension - ≥180, Isolated systolic hypertension - ≥140.
  Diastolic BP (measured in mmHg): Optimal - <80, Normal - 80 - 84, High normal - 85 - 89, Grade 1 hypertension - 90 - 99, Grade 2 hypertension - 100 - 109, Grade 3 hypertension - ≥110, Isolated systolic hypertension - < 90.
To assess the safety and tolerability of VL-SE-01 on Pulse Rate. | Day 0, Day 90, Day 180 and Day 195
  Vitals signs measures basic functions of the body. In this case Heart rate [also known as Pulse rate (PR)] will be measured.
  Pulse rate will be measured by palpatory method by counting the number of beats in 30 seconds.
  Normal Pulse rate: 60 - 100 beats per minute (bpm) Bradycardia: < 60 bpm Tachycardia: > 100 bpm
To assess the safety and tolerability of VL-SE-01 using Electrocardiogram. | Day 0, Day 90, Day 180 and Day 195
  The electrocardiograph is a device that picks up electrical activity originating in the heart from the surface of the body for clinical diagnosis of cardiac function. The following parameters will be considered for the study:
  The QT interval is the time from the beginning of the QRS complex, representing ventricular depolarization, to the end of the T wave, resulting from ventricular repolarization. In general, the normal QT interval is below 400 to 440 milliseconds (ms), or 0.4 to 0.44 seconds. Women have a longer QT interval than men.
  The corrected QT interval (QTc) estimates the QT interval at a standard heart rate of 60 bpm. Normal values for the QTc range from 350 to 450 ms for adult men and from 360 to 460 ms for adult women; however, 10%-20% of otherwise healthy persons may have QTc values outside this range.
  The PR interval is the time from the beginning of the P wave (atrial depolarization) to the beginning of the QRS complex (ventricular depolarization). The normal
To assess the safety and tolerability of VL-SE-01 using Treatment emergent Adverse Events (TEAEs). | Day 0, Day 90, Day 180 and Day 195
  The number and percent of research participants reporting AEs will be tabulated by intervention group and will be compared between the groups.
To evaluate the efficacy of VL-SE-01 on the basis of Incidence of gastrointestinal dysfunction using Structured Assessment of Gastrointestinal Symptoms (SAGIS) questionnaire. | Day 0, Day 90, and Day 180
  SAGIS is a suitable questionnaire to assess gastrointestinal complaints like Decreased appetite, Diarrhea, Weight decreased, Gastroenteritis Abdominal pain, discomfort etc.
  It consists of 22 items as well as two open questions asking for the participant's most and second most important clinical problem. Q1 to Q22 are summed together to give a total symptom burden score. The total symptoms burden score can range from 0 to 88.The number of items between Q1 and Q22 that are scored severe (3) or very severe (4) are added together. The global impact score can range from 0 to 22.
To evaluate the efficacy of VL-SE-01 on the basis of Sleep quality using the PSQI questionnaire | Day 0, Day 90, and Day 180
  The questions relate to a person's usual sleep habits during the past month. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). All the seven component scores are to be added together for calculating the Global PSQI Score. Higher scores indicate worse sleep quality.
To evaluate the efficacy of VL-SE-01 on the basis of Insomnia using Insomnia Severity Index (ISI) | Day 0, Day 90, and Day 180
  The questionnaire evaluates the sleep quality in last two weeks. The seven answers are added up to the total score.The scores of 0-7 determines no clinically significant insomnia, 8-14 determines sub threshold insomnia, 15-21 has moderate severity which determines clinical insomnia and lastly 22-28 has severe insomnia.
To evaluate the efficacy of VL-SE-01 on the basis of Fatigue will be assessed using fatigue severity scale (FSS) | Day 0, Day 90, and Day 180
  The FSS is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Grading of each item ranges from 1 to 7, where 1 indicates strong disagreement and 7 indicates strong agreement, and the final score represents the mean value of the 9 items.
  A visual analogue scale is also included with the scale in which the respondents will be asked to denote the severity of their fatigue at the present moment by placing a mark on a line extending from "no fatigue" to "fatigue as bad as could be." Higher scores on the scale are indicative of more severe fatigue
To evaluate the efficacy of VL-SE-01 on the basis of Stress response as assessed by Perceived Stress Scale (PSS). | Day 0, Day 90, and Day 180
  The questions in this scale ask about feelings and thoughts of an individual during the last month.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress
To evaluate the efficacy of VL-SE-01 on the basis of Menstrual cycle regularity. | Day 0, Day 90, and Day 180
  A diary will be provided to the participant to record their monthly menstruation period start date and stop date. The average length of a menstrual cycle is of 28 days, however it varies for every female.
To evaluate the efficacy of VL-SE-01 on the basis of Plasma levels of CBD and its metabolites [7-Carboxy-cannabidiol (7-COOH-CBD) and 7-Hydroxy-cannabidiol (7-OH-CBD)] | 0 hour, 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours at Day 0, Day 90, Day 180
  This will be conducted in 15 participants only in each group except placebo.

CONTACTS AND LOCATIONS:
Locations (6):
- India (6):
  - Shivam Hospital, Dombivali, Maharashtra
  - Dhanwantri Hospital, Pune, Maharashtra
  - Vedant Multispeciality Hospital, Pune, Maharashtra
  - Punawale Hospital, Pune, Maharashtra
  - Vishwaraj Hospital, Pune, Maharashtra
  - Shree Ashirwad Hospital, Thane, Maharashtra

IPD SHARING:
Plan to Share IPD: No